CLINICAL TRIAL: NCT06654180
Title: A Comparison of Myopia Control Efficacy in Children With Orthokeratology, Defocus Incorporated Multiple Segment (DIMS) Spectacles, Defocus Incorporated Soft Contact (DISK) Lenses, and Single-vision Spectacles for 12 Months
Brief Title: Comparing Myopia Control Efficacy in Children With 4 Methods: Orthokeratology, DIMS, DISK, and SVS.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaikai QIU (Other)
Collaborators: Ningbo Eye Hospital (Other)
Responsible Party: Sponsor-Investigator, Kaikai QIU, Researcher, Fuzhou Southeast Institute of Visual Ophthalmology
Organization: Fuzhou Southeast Institute of Visual Ophthalmology (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Southeast Eye Institute; MR-33-22-012252 (Registry Identifier: Research Committee of China Medical Institute)
Record Dates: First submitted 2024-10-16; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Myopia
Keywords: Myopia; Children
MeSH Terms: conditions — Myopia | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Orthokeratology (Active Comparator): To wear Orthokeratology at night to slow down progressing myopia
  Interventions: Device: Orthokeratology
- defocus-incorporated multiple segment lenses (DIMS) spectacles (Experimental): To wear defocus-incorporated multiple segment lenses (DIMS) spectacles at daytime
  Interventions: Device: defocus-incorporated multiple segment lenses (DIMS) spectacles
- defocus incorporated soft contact (DISK) lenses (Experimental): To wear defocus incorporated soft contact (DISK) lenses at daytime
  Interventions: Device: DISK
- single-vision spectacles (SVS) (Placebo Comparator): To wear SVS at daytime and at night before sleep
  Interventions: Device: Single-focus spectacles

INTERVENTIONS:
Device: Orthokeratology — Orthokeratology is to a rigid contact lens with reverse design to flat the central cornea to correct the myopia, which is to use at night during sleep; DIMS and SVS are both spectacles to wear at daytime; DIMS has many tiny lenses at peripheral of the big lenses to make the peripheral retina myopic defocus during the daytime; SVS has only one focus while DIMS has many focuses made by the tiny segments lenses around the peripheral vision fields; DISK is a soft contact lens with peripheral myopic power design to make the myopic eyes defocus at peripheral during the daytime.
  Other Names: DIMS; DISK; SVS
  Arms: Orthokeratology
Device: defocus-incorporated multiple segment lenses (DIMS) spectacles — It is the special lenses with peripheral lots of tiny segments of plus lenses around the center
  Arms: defocus-incorporated multiple segment lenses (DIMS) spectacles
Device: DISK — SVS
  Arms: defocus incorporated soft contact (DISK) lenses
Device: Single-focus spectacles — Myopic Glasses with mono-focus in each eye
  Arms: single-vision spectacles (SVS)

SUMMARY:
The goal of this clinical trial is to learn if 3 optical interventions（DIMS, DISC and orthokeratology) to control myopia have different efficacy to slow myopia progression in children when the control is single focus spectacles(SVS). It will also learn about the safety of all 4 interventions. The main questions it aims to answer are:

Does orthokeratology slows the progressing myopia more significant than the DIMS or DISK? What medical problems do participants have when taking orthokeratology, DIMS and DISK? Researchers will compare all the 3 interventions to a placebo (SVS) to see if 3 interventions has significant difference in slow the axial length elongation as well as the refraction changes.

Participants will:

Take orthokeratology, DIMS, DISK or SVS every day for 12 months Visit the clinic once every 3 months for checkups and tests.

DETAILED DESCRIPTION:
orthokeratology and DISK are contact lenses, while DIMS and SVS are spectacles.

ELIGIBILITY:
Inclusion Criteria:

* Must agree to participate in the study
* Must have cycloplegic refraction with spherical equivalent refractive (SER)

  * - 2.00 D ~ - 5.00 D (including the boundary values)
* Clinical diagnosis of astigmatism was ≤ 1.00D
* Must be able to have corrected visual acuity ≤ 0.00 logMAR of either eye
* Must be able to wear either of SVS/DIMS/DISC/Orthokeratology lenses and kept the same intervention for 12 month
* Must have the front cornea curve value between 41.00D~44.00D
* Must have axial length of the study eye between 23.00mm and 25.00mm at baseline

Exclusion Criteria:

* Dry eye
* keratitis
* Conjunctivitis
* Clinical diagnosis of entropion
* Clinical diagnosis of glaucoma
* Clinical diagnosis of retinal lesions
* Clinical diagnosis of amblyopia
* Clinical diagnosis of optic media lesions (e.g., central thick corneal scars, cataract)
* Clinical diagnosis of optic nerve dysfunction
* Have medical history of atropine eyedrops (including 1% high concentration , 0.05%, 0.01% or other low concentration)
* Have history of wearing peripheral defocus spectacles
* Have history of wearing duo-focal soft contact lenses
* Unable to follow up
* Investigators consider to be not eligible.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — All the genders are welcome to join the clinical trials. While those who is self-identified genders are eligible to participate while the record is not male or female.
Enrollment: 100 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-10 (Estimated)

PRIMARY OUTCOMES:
Changes of axial length for 12-month (mm) | 12 months
  The ocular axial length change at follow-up of 12-month from baseline with IOLmaster 500（IOLMaster 500, Carl Zeiss Meditec AG, Germany) in the unit of millimetre

SECONDARY OUTCOMES:
Changes of Spherical Equivalence Refraction (D) | 12 months
  Changes of SER at 12-Month follow-up with cycloplegic refraction (Diopter, D) with the auto refractometer (Topcon KR-800, Topcon Corporation, Tokyo, Japan)
Dropout rate (%) | 12 months
  The dropout rate of each group with the percentage (%) record by the formula =the dropout number versus total number of the each group *100%.
Changes of ocular axial length at follow-up of 3 months (mm) | 3 months
  Changes of ocular axial length at follow-up of 3 month from baseline with the IOLmaster 500(millimetre, mm)
Changes of ocular axial length at follow-up of 6 months (mm) | 6 months
  Changes of ocular axial length at follow-up of 6 month from baseline with the IOLmaster 500(millimetre, mm)
Changes of ocular axial length at follow-up of 9 months (mm) | 9 months
  Changes of ocular axial length at follow-up of 9 month from baseline with the IOLmaster 500(millimetre, mm)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Ningbo Eye Hospital, Ningbo, Zhejiang
  - Optometry department, Ningbo Eye Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No
The explanation why IPD will not be shared is that almost all the data to be obtained is on another clinic center with another external site. The data is confidential to obtain to outside system with complete details.